CLINICAL TRIAL: NCT02004860
Title: Phase 3 : Tacrolimus Ointment Interest (PROTOPIC ®) in the Maintenance Treatment of Severe Seborrheic Dermatitis on Adult Face
Brief Title: Tacrolimus Ointment Interest (PROTOPIC ®) in the Maintenance Treatment of Severe Seborrheic Dermatitis
Acronym: Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011/104/HP; 2011-004186-32 (EudraCT Number)
Record Dates: First submitted 2013-08-26; First posted 2013-12-09 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Severe Seborrheic Dermatitis
Keywords: local immunosuppressive; Maintenance therapy
MeSH Terms: conditions — Dermatitis, Seborrheic | interventions — Tacrolimus; Ciclopirox

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Protopic Arm (Experimental): Protopic® 0.1% ointment - 2 applications per week for 6 months
  Interventions: Drug: Protopic (R)
- Mycoster Arm (Active Comparator): 2 applications per week for 6 months
  Interventions: Drug: Mycoster (R)

INTERVENTIONS:
Drug: Protopic (R) — Protopic® 0.1% ointment - 2 applications per week for 6 months
  Other Names: Tacrolimus
  Arms: Protopic Arm
Drug: Mycoster (R) — Mycoster 1% - 2 applications per week for 6 months
  Other Names: Ciclopirox olamine
  Arms: Mycoster Arm

SUMMARY:
Seborrheic dermatitis is a chronic inflammatory dermatological disease, evolving by relapses, affecting mainly the face and scalp. It would be important to have a maintenance treatment for severe forms of seborrheic dermatitis witch is both effective and relatively well tolerated to reduce the frequency of relapses, prolong remissions obtained after attack treatment and reduce the use of topical steroids.

ELIGIBILITY:
Inclusion Criteria:

* in Phase 1: Attack Treatment (open)

  1. over the age of eighteen patient,
  2. Seborrheic dermatitis Severe,
  3. participation with an informed consent,
  4. Women of childbearing age in effective contraception for the duration of the study or postmenopausal women.
* in Phase 2: Phase 2: "Randomization" (blind)

  1. Patient achieved a complete or almost complete clinical remission after the initial treatment,
  2. known immunodeficiency (HIV patient receiving chemotherapy) or immunosuppressive therapy or biotherapy,
  3. patient taking regular systemic corticosteroids at a dose> 20 mg / day
  4. erythematous lesions with topography other than the face and evocative scalp psoriasis (elbows, knees ...), by referring to the possibility that the facial lesions correspond to lesions sebopsoriasis,
  5. woman pregnant, nursing or in childbearing potential without effective contraception,
  6. man wishing to have a child during the study period,
  7. Ultra Violet (UV) phototherapy or usual realization of UV sessions aesthetic purposes,
  8. Seborrheic dermatitis symptomatic of an underlying disease known or revealing
  9. history of cancer or lymphoma,
  10. progressive cancer or lymphoma,
  11. Seborrheic dermatitis exclusively affecting the scalp,
  12. known allergy to one-component products study ,
  13. malnourished patient or sick history of chronic pancreatitis by a suspect to deficiency dermatitis,
  14. participation in a clinical trial on the Seborrheic dermatitis in the previous 90 days,
  15. patient with lesions considered potentially malignant or pre-cancerous,
  16. patient with abnormal skin barrier.

Exclusion Criteria:

* in Phase 1: Attack Treatment (open)

  1) Patient had already been treated with Protopic ® for Seborrheic Dermatitis,
* Phase 2: "Randomization" (blind) 1) Patient with no complete or almost complete clinical remission after the initial treatment,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-01; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
duration of the maintenance of complete or almost complete clinical remission | 18 months after inclusion (Visit (V) 4 last visit)
  The primary endpoint will be the duration of the maintenance of complete or almost complete clinical remission obtained after the initial treatment. This period is defined as the time from randomization to the first occurrence of relapse noted by the dermatologist.

SECONDARY OUTCOMES:
Tolerance of 2 treatments | between 10 days and 18 months after inclusion (V3 (Day (D)10 to D180)), 30 days after inclusion (Visit D30), after 90 days after inclusion (D90) and after 120 days after inclusion (D120) and 180 days after inclusion (Visit V4)
  Tolerance of 2 treatments Mycoster (R) and Protocopic (R)
Number of Relapses | 180 days after inclusion (Visit V4)
  Number of Relapses requiring the resumption of topical corticosteroid treatment,
Cumulative amount of corticosteroids applied | between 10 days and 18 months after inclusion (V3 (D10 to D180)), 30 days after inclusion (Visit D30), after 90 days after inclusion (D90) and after 120 days after inclusion (D120) and 180 days after inclusion (Visit V4)
  Cumulative amount of corticosteroids applied by the patients during the study period to control their outbreaks
quality of life of patients | Inclusion (visit D0) and Last visit 180 days after inclusion (Visit D180)
  quality of life of patients

CONTACTS AND LOCATIONS:
Overall Officials: Pascal JOLY, Professor, Study Director — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France